CLINICAL TRIAL: NCT00758680
Title: A Multiple Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-1006.
Brief Title: A Multiple-Dose Study of MK-1006 (MK-1006-004)(TERMINATED)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1006-004; 2008_550
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- MK-1006 20 mg Once Daily (Panel A) (Experimental): After a 2-week run-in/wash-off period, participants received single daily doses (q.d.) of 20 mg MK-1006 over a 10-day multiple-dosing period while remaining domiciled in the Clinical Research Unit (CRU).
  Interventions: Drug: MK-1006
- MK-1006 40 mg Once Daily (Panel B) (Experimental): After a 2-week run-in/wash-off period, participants received single daily doses of 40 mg MK-1006 over a 10-day multiple-dosing period while remaining domiciled in the CRU.
  Interventions: Drug: MK-1006
- MK-1006 80 mg Once Daily (Panel C) (Experimental): After a 2-week run-in/wash-off period, participants received single daily doses of 80 mg MK-1006 over a 10-day multiple-dosing period while remaining domiciled in the CRU.
  Interventions: Drug: MK-1006
- MK-1006 120 mg Once Daily (Panel D) (Experimental): After a 2-week run-in/wash-off period, participants received single daily doses of 120 mg MK-1006 over a 10-day multiple-dosing period while remaining domiciled in the CRU.
  Interventions: Drug: MK-1006
- MK-1006 20 mg Twice Daily (Panel E) (Experimental): After a 2-week run-in/wash-off period, participants received twice-daily doses (b.i.d.) of 120 mg MK-1006 over a 10-day multiple-dosing period while remaining domiciled in the CRU.
  Interventions: Drug: MK-1006
- MK-1006 30 mg Twice Daily (Panel F) (Experimental): After a 2-week run-in/wash-off period, participants received twice-daily doses of 30 mg MK-1006 over a 10-day multiple-dosing period while remaining domiciled in the CRU.
  Interventions: Drug: MK-1006
- MK-1006 50 mg Twice Daily (Panel G) (Experimental): After a 2-week run-in/wash-off period, participants received twice-daily doses of 50 mg MK-1006 over a 10-day multiple-dosing period while remaining domiciled in the CRU.
  Interventions: Drug: MK-1006
- MK-1006 120 mg Once Daily Outpatient (Panel H) (Experimental): After a 2-week run-in/wash-off period, participants received single daily doses of 120 mg MK-1006 over a 7-day multiple-dosing period while remaining domiciled in the CRU. Participants were then discharged from the CRU and continued daily dosing of MK-1006 for an additional 21 days as outpatients.
  Interventions: Drug: MK-1006
- MK-1006 50 mg Twice Daily Outpatient (Panel I) (Experimental): After a 2-week run-in/wash-off period, participants received twice-daily doses of 50 mg MK-1006 over a 7-day multiple-dosing period while remaining domiciled in the CRU. Participants were then discharged from the CRU and continued daily dosing of MK-1006 for an additional 21 days as outpatients.
  Interventions: Drug: MK-1006
- Placebo (Placebo Comparator): After a 2-week run-in/wash-off period, participants received dose-matched placebo to MK-1006 over a multiple-dosing period while remaining domiciled in the CRU.
  Interventions: Drug: Comparator: Placebo comparator

INTERVENTIONS:
Drug: MK-1006 — MK-1006 capsules (10 mg and 20 mg) administered orally from 20 mg to 120 mg per dose over a multiple dosing period.
  Arms: MK-1006 120 mg Once Daily (Panel D); MK-1006 120 mg Once Daily Outpatient (Panel H); MK-1006 20 mg Once Daily (Panel A); MK-1006 20 mg Twice Daily (Panel E); MK-1006 30 mg Twice Daily (Panel F); MK-1006 40 mg Once Daily (Panel B); MK-1006 50 mg Twice Daily (Panel G); MK-1006 50 mg Twice Daily Outpatient (Panel I); MK-1006 80 mg Once Daily (Panel C)
Drug: Comparator: Placebo comparator — Dose-matched MK-1006 placebo capsules (1 mg, 10 mg and 20 mg) administered orally over a multiple dosing period.
  Arms: Placebo

SUMMARY:
This study will asses the safety, tolerability, multiple-dose pharmacokinetics and pharmacodynamics of MK1006 in participants with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a BMI less than or equal to 42 kg/m^2 at the screening visit
* Participant has been diagnosed with Type 2 Diabetes that is being treated either by diet and exercise alone or by single or combination oral anti-hyperglycemic medications
* Participant is willing to follow a diet containing approximately 50% carbohydrates, 20% protein, and 30% fat during the study
* Participant is a nonsmoker and has not used nicotine containing products for ~ 6 months before start of study

Exclusion Criteria:

* Participant must not be treated with three or more oral anti-hyperglycemic medications, insulin, or PPAR-gamma agonists
* Participant has a history of stroke, chronic seizures, or a major neurological disorder
* Participant has had an eye infection or other inflammatory eye condition within 2 weeks of first dose of study drug
* Participant has glaucoma or is blind
* Participant has a condition known to be related to cataract development
* Participant has had or will have incisional eye surgery within 6 months before screening or has had laser surgery (other than Lasik) within 3 months of screening
* Participant has a history of type 1 diabetes or ketoacidosis
* Participant cannot stop taking certain current medications during the study
* Participant consumes greater than 3 alcoholic beverages per day
* Participant consumes more than 6 servings of caffeinated beverages per day (1 serving is ~ 120 mg caffeine)
* Participant has a history of significant multiple or severe allergies or has had a reaction to or is intolerant of prescription/non-prescription drugs or food
* Participant uses recreational drugs or has had a history of drug abuse within 6 months of start of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-1006 20 mg Once Daily (Panel A) | MK-1006 40 mg Once Daily (Panel B) | MK-1006 80 mg Once Daily (Panel C) | MK-1006 120 mg Once Daily (Panel D) | MK-1006 20 mg Twice Daily (Panel E) | MK-1006 30 mg Twice Daily (Panel F) | MK-1006 50 mg Twice Daily (Panel G) | MK-1006 120 mg Once Daily Outpatient (Panel H) | MK-1006 50 mg Twice Daily Outpatient (Panel I) | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 20 | 20 | 29
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 19 | 18 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Laboratory Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treated Participants: After a 2-week run-in/wash-off period, participants received doses of MK-1006 or matching placebo over a multiple-dosing period while remaining domiciled in the Clinical Research Unit (CRU).
Arm/Group | All Treated Participants
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) On Study
Description: An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the study treatment, was also an adverse event.
Time Frame: From Day 1 through the end of poststudy period (up to Day 25)
Population: All Participants as Treated (APaT); All participants who received at least one dose of the investigational drug
Measure: Number; unit: participants
Arm/Group | MK-1006 20 mg Once Daily (Panel A) | MK-1006 40 mg Once Daily (Panel B) | MK-1006 80 mg Once Daily (Panel C) | MK-1006 120 mg Once Daily (Panel D) | MK-1006 20 mg Twice Daily (Panel E) | MK-1006 30 mg Twice Daily (Panel F) | MK-1006 50 mg Twice Daily (Panel G) | MK-1006 120 mg Once Daily Outpatient (Panel H) | MK-1006 50 mg Twice Daily Outpatient (Panel I) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 20 | 20 | 29
participants | 1 | 1 | 4 | 5 | 4 | 4 | 6 | 15 | 16 | 22

2. Secondary Outcome: Least Squares Mean Change From Baseline in 24-Hour Weighted Mean Glucose (WMG)
Description: Plasma glucose concentration was determined using a glucometer and measured before drug was given to establish a baseline fasting plasma glucose concentration. Plasma glucose concentrations were then measured every ~30 minutes over a 24 hour period after the Day 1 dose (First Dosing Day) and after the Day 10 dose (Last Dosing Day) to obtain a weighted mean average value for Day 1 and for Day 10. Results were expressed as the change from baseline to the Day 1 weighted average (First Dosing Day), and as the change from baseline to the Day 10 weighted average (Last Dosing Day).
Time Frame: Day -1 (pre-dose baseline), Day 1 (First Dosing Day), Day 10 (Last Dosing Day)
Population: Per-Protocol Population; subset of participants who complied with the protocol sufficiently in terms of considerations as exposure to treatment, availability of measurements and absence of major protocol violations.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-1006 20 mg Once Daily (Panel A) | MK-1006 40 mg Once Daily (Panel B) | MK-1006 80 mg Once Daily (Panel C) | MK-1006 120 mg Once Daily (Panel D) | MK-1006 20 mg Twice Daily (Panel E) | MK-1006 30 mg Twice Daily (Panel F) | MK-1006 50 mg Twice Daily (Panel G) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
mg/dL
  First Dosing Day | -5.3 (11.3) | -19.3 (15.1) | -43.8 (10.1) | -41.5 (6.3) | -20.7 (10.3) | -26.4 (20.3) | -42.5 (18.6) | 5.3 (11.1)
  Last Dosing Day | 3.5 (40.1) | 0.8 (73.8) | -66.9 (20.3) | -7.4 (51.4) | -40.3 (8.7) | -30.7 (30.8) | -62.1 (18.8) | 30.2 (40.6)
Statistical Analysis 1: Comparison: MK-1006 120 mg Once Daily (Panel D) vs Placebo; Test type: Superiority or Other; p = 0.015, Mixed Effect Model; LS Mean Difference on Last Dosing Day = 37.63, 95% CI 2-sided [12.58 to 62.68]
Statistical Analysis 2: Comparison: MK-1006 50 mg Twice Daily (Panel G) vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Effect Model; LS Mean Difference on Last Dosing Day = 92.30, 95% CI 2-sided [67.56 to 117.04]

3. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 1
Time Frame: From Day 1 through the end of poststudy period (up to Day 25)
Population: All Participants as Treated (APaT); All participants who received at least one dose of the investigational drug
Measure: Number; unit: participants
Arm/Group | MK-1006 20 mg Once Daily (Panel A) | MK-1006 40 mg Once Daily (Panel B) | MK-1006 80 mg Once Daily (Panel C) | MK-1006 120 mg Once Daily (Panel D) | MK-1006 20 mg Twice Daily (Panel E) | MK-1006 30 mg Twice Daily (Panel F) | MK-1006 50 mg Twice Daily (Panel G) | MK-1006 120 mg Once Daily Outpatient (Panel H) | MK-1006 50 mg Twice Daily Outpatient (Panel I) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 20 | 20 | 29
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

ADVERSE EVENTS:
Arm/Group | MK-1006 20 mg Once Daily (Panel A) | MK-1006 40 mg Once Daily (Panel B) | MK-1006 80 mg Once Daily (Panel C) | MK-1006 120 mg Once Daily (Panel D) | MK-1006 20 mg Twice Daily (Panel E) | MK-1006 30 mg Twice Daily (Panel F) | MK-1006 50 mg Twice Daily (Panel G) | MK-1006 120 mg Once Daily Outpatient (Panel H) | MK-1006 50 mg Twice Daily Outpatient (Panel I) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 1/20 | 0/20 | 1/29
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 4/6 | 5/6 | 2/6 | 4/6 | 6/7 | 15/20 | 16/20 | 22/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1006 20 mg Once Daily (Panel A) (N=6) | MK-1006 40 mg Once Daily (Panel B) (N=6) | MK-1006 80 mg Once Daily (Panel C) (N=6) | MK-1006 120 mg Once Daily (Panel D) (N=6) | MK-1006 20 mg Twice Daily (Panel E) (N=6) | MK-1006 30 mg Twice Daily (Panel F) (N=6) | MK-1006 50 mg Twice Daily (Panel G) (N=7) | MK-1006 120 mg Once Daily Outpatient (Panel H) (N=20) | MK-1006 50 mg Twice Daily Outpatient (Panel I) (N=20) | Placebo (N=29)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-1006 20 mg Once Daily (Panel A) (N=6) | MK-1006 40 mg Once Daily (Panel B) (N=6) | MK-1006 80 mg Once Daily (Panel C) (N=6) | MK-1006 120 mg Once Daily (Panel D) (N=6) | MK-1006 20 mg Twice Daily (Panel E) (N=6) | MK-1006 30 mg Twice Daily (Panel F) (N=6) | MK-1006 50 mg Twice Daily (Panel G) (N=7) | MK-1006 120 mg Once Daily Outpatient (Panel H) (N=20) | MK-1006 50 mg Twice Daily Outpatient (Panel I) (N=20) | Placebo (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lenticular Opacities (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Application Site Irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver Disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Glucose Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 5 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 3 | 2 | 0 | 6 | 3 | 5 | 4
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Coldness (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.